CLINICAL TRIAL: NCT00135187
Title: A Pilot Study of Combination Therapy With VELCADE, Doxil, and Dexamethasone (VDd) in Multiple Myeloma
Brief Title: Study of Combination Therapy With VELCADE, Doxil, and Dexamethasone (VDd) in Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Andrzej J. Jakubowiak, MD, PhD, University of Michigan Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004.003; Legacy 2004-419 (Other: University of Michigan IRBMED); NCT00670085 (obsolete NCT alias)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; liposomal doxorubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: VELCADE — VELCADE will be used biweekly at 1.3 mg/m2 during week 1 and 2 on (days
  1, 4, 8, and 11) followed by a 1-week break.
Drug: Doxil — Doxil will be administered at 30 mg/m2 IV on day 4
Drug: Dexamethasone — Dexamethasone at 40 mg during the first cycle and 20 mg during cycles 2-6 po or IV daily on days of VELCADE and day after VELCADE (i.e. days 1, 2, 4, 5, 8, 9, 11, 12). The patient will be treated for six 3-week cycles followed by three 5-week maintenance cycles.

SUMMARY:
Patients are being asked to take part in this research study because they have multiple myeloma which has relapsed after (come back), or is refractory to (unaffected by), initial therapy.

For patients who have relapsed or are refractory to therapy, there is no agreed upon standard treatment. Treatment options include chemotherapy and, for some patients, bone marrow transplants. None of the available treatments are curative and investigators are continually looking for more effective treatments. This study involves treatment with a new combination of standard drugs: VELCADE, Doxil, and Dexamethasone. Preliminary results from a study using a combination of VELCADE with Doxil showed high response rates (disease reduction). Two other studies showed that an addition of Dexamethasone to VELCADE in patients not responding to VELCADE alone improved response rate. The proposed combination of all three drugs may improve efficacy and response.

VELCADE is approved by the Food and Drug Administration (FDA) for use in multiple myeloma. Doxil is not approved for use in multiple myeloma but is an approved drug for use in patients with some other cancers. Several published clinical trials provide evidence that Doxil is an active agent in multiple myeloma and it is used in treatment combinations for multiple myeloma in general practice. Dexamethasone is approved for use in multiple myeloma. The combination of all three drugs is experimental (not FDA approved).

The goals of this study are to determine if this new combination therapy with VELCADE, Doxil and Dexamethasone is an effective treatment, and also to determine the side effects that occur when this combination treatment is given.

DETAILED DESCRIPTION:
Multiple myeloma remains a non-curable disease. Combination therapies such as VAD have been effective, with partial response rates in ~40-60% range and tolerable toxicity. A recent study showed that substituting Doxil for Doxorubicin in a regimen similar to VAD (DVd) resulted in an improved toxicity profile and similar efficacy. The most active agents in VAD (and presumably in DVd) are Doxorubicin (or Doxil) and Dexamethasone, while Vincristine adds little, if at all to the efficacy of these regimen(s). One of the new active agents in multiple myeloma is VELCADE (bortezomib, formerly known as VELCADE). This molecule has a novel mechanism of action by specifically inhibiting the proteasome. A recently reported Phase II trial showed that VELCADE as a single agent induced at least minimal responses (i.e. > 25% reduction in monoclonal protein) in 35% of patients and at least a stabilization of the disease in 59% of patients with relapsed/refractory multiple myeloma using strict SWOG criteria. An additional 18% responded when Dexamethasone was added to VELCADE. Pre-clinical observations showed that the addition of VELCADE to other chemotherapeutic agents, such as doxorubicin, enhances cytotoxicity of multiple myeloma cells. Preliminary results from Phase I study of combination of VELCADE with Doxil showed 60% response rate (i.e. > partial response) with acceptable toxicity. In this study we propose to combine three active agents, i.e. Doxil, Dexamethasone (two most active agents from DVd), and VELCADE. The ultimate goal is to show that this combination of drugs is more efficacious than VAD or VELCADE with either Dexamethasone or Doxil and without additional toxicity.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* An Institutional Review Board (IRB)-approved signed informed consent
* Patient is, in the investigator's opinion, willing and able to comply with the protocol requirements
* Age greater than or equal to 18 years
* Female patient is either postmenopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e. hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male patient agrees to use an acceptable method of contraception for the duration of the study
* Expected survival greater than or equal to 3 months
* Pre-study Karnofsky performance status > 60%
* Histologic confirmation of multiple myeloma
* Patient was previously diagnosed with stage II or III multiple myeloma based on standard criteria and currently requires second or higher line therapy because of progression of disease (PD), defined as a 25% increase in M-protein; development of new or worsening of existing lytic lesions or soft tissue plasmacytomas; or hypercalcemia (> 11.5 mg/dl); or relapse from complete response (CR) or because of refractory disease, defined as less than minimal response (MR) after 2 cycles of the most recent treatment, including first line of therapy.
* Patients with measurable disease defined as: serum monoclonal protein greater than 1 g/dl for IgG type and greater than 0.5 g/dl for IgA type, and, where applicable, greater than 0.2 g/24 hour urine light chain excretion.
* Patients with oligosecretory or nonsecretory myeloma will be eligible if measurable disease can be established, such as measurable soft tissue plasmacytoma greater than 2 cm, by either physical examination and/or applicable radiographs (i.e. magnetic resonance imaging [MRI], computed tomography [CT]-scan) and/or bone marrow involvement greater than 20%.
* Patients refractory or relapsing after treatment with any one or two of the agents used in this protocol will be allowed.
* Prior radiation therapy will be allowed but radiation therapy must be completed 2 weeks prior to registration.
* Left ventricular ejection fraction (LVEF) > 50% by multiple-gated acquisition (MUGA) or echocardiogram (ECHO)
* Patients previously on investigational drugs if no long-term toxicity is expected, and the patients have been off the drugs for one or more weeks
* Patient has received less than 250 mg/m2 cumulative dose of doxorubicin or equivalent.
* Patient has the following laboratory values at and within 14 days before Baseline (Day 1 of Cycle 1, before study drug administration):

  * Platelet count > 50 x 10^9/L without transfusion support within 7 days before the laboratory test (> 30 x 10^9/L if significant bone marrow [BM] involvement is present);
  * Hemoglobin > 7.5 x 10^9/L, without transfusion support within 7 days before the laboratory test;
  * Absolute neutrophil count (ANC) > 1.0 x 10^9/L, without the use of colony stimulating factors;
  * Corrected serum calcium < 14 mg/dl (3.5 mmol/L);
  * Aspartate transaminase (AST): < 2.5 x upper limit of normal (ULN);
  * Alanine transaminase (ALT): < 2.5 x ULN;
  * Alkaline phosphatase: <1.5 x the ULN;
  * Total bilirubin: < 1.5 x the ULN; and
  * Calculated or measured creatinine clearance: > 20 mL/minute.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Patient had major surgery within 3 weeks before enrollment.
* Patient had a myocardial infarction within 6 months of enrollment or clinical evidence of congestive heart failure.
* Patient is known to be human immunodeficiency virus (HIV)-positive (patients assessed to be at risk should be tested).
* Patient is known to be hepatitis B surface antigen-positive or has known active hepatitis C infection (patients assessed by the investigator to be at risk should be tested)
* Patient has >= Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has hypersensitivity to bortezomib, boron or mannitol, or other study drugs.
* Serious nonmalignant disease, including uncontrolled diabetes mellitus (DM) or hypertension (HTN), or infection which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2006-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Estimate an overall response rate to combination therapy with VELCADE, Doxil, and Dexamethasone, defined as at least partial response (PR), i.e. > 50% reduction in serum monoclonal protein and/or >90% reduction in Bence-Jones protein by EBMT criteria. | 6 months
  Multiple myeloma remains a non-curable disease. Combination therapies such as VAD have been effective, with partial response rates in ~40-60% range and tolerable toxicity. The purpose of this study is to see if this combination is more effective

SECONDARY OUTCOMES:
Estimate a rate of complete response (CR), very good partial response (VGPR, >90% reduction in serum monoclonal protein), minimal response (MR, >25% and <50% reduction in monoclonal) | 6 months
Estimate the duration of response, progression-free survival, overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej J Jakubowiak, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States